CLINICAL TRIAL: NCT06303466
Title: Real World Evidence Study of Danish Fabry Patients: a >20- Year Longitudinal Retrospective Analysis of Prospectively Collected Data.
Brief Title: Real World Evidence Study of Danish Fabry Patients
Acronym: RWE-FABRY
Status: Active, not recruiting | Type: Observational
Sponsor: Caroline Michaela Kistorp (Other)
Collaborators: Amicus Therapeutics (Industry); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Caroline Michaela Kistorp, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: R-23053109
Record Dates: First submitted 2024-02-14; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Fabry Disease
Keywords: Cardiovascular Diseases; Renal Disease; Cerebrovascular disease
MeSH Terms: conditions — Fabry Disease; Cardiovascular Diseases; Kidney Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and urine samples collected over the last 20+ years as part of routine monitoring of patients with Fabry Disease by the Danish National Fabry Center at Rigshospitalet, Copenhagen University Hospital, Denmark.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Danish Fabry Patients: Patients with a genetically-verified diagnosis of Fabry Disease.

SUMMARY:
Fabry is a rare X-linked metabolic lysosomal disorder caused by deficiency in the enzyme α-galactosidase A (alpha-Gal A) by mutations in the GLA gene, encoding the alpha-Gal A enzyme, which catalyses glycosphingolipids, namely globotriaosylceramide (Gb3). Reduced or absent alpha-Gal A activity leads to accumulation of Gb3 in various organs as well as cellular dysfunction and inflammation causing phsyical symptoms and eventual organ failure. Treatment has been available since 2001 for Fabry patients - first enzyme replacement therapy and since 2016, an oral chaperone therapy, Migalastat. Although the initial trials of Migalastat had some both short and extended outcome treatment comparisons, the overall evidence of clinical efficacy is based on too small numbers considering the heterogeneity of the Fabry patient population as well as the very slow progression of the disease. Though the body of real-world evidence is growing, there is a need for more publications of real-world long-term data on clinical outcomes with a focus on treatment with Migalastat.

Research Question:

Is the incidence and prevalence of Fabry associated clinical events (FACEs) (cardiac, renal, and cerebrovascular) associated with sex, genotype, phenotype at time of diagnosis, biomarkers, and Fabry specific therapy?

Objectives:

* To investigate time to first Fabry associated clinical events (FACE) (cardiac, renal, and cerebrovascular) with particular focus on Migalastat clinical outcomes and treatment outcomes preceding Migalastat therapy.
* To investigate the incidence and prevalence of FACEs with respect to Fabry specific treatment, Migalastat, ERT or no treatment.
* To describe FACEs in accordance with different geno- and phenotypic groups.
* To investigate the incidence and time to a first fatal or non-fatal cardiac, renal, and cerebrovascular clinical event, separated by each category.

Primary outcomes - Time to first FACE (cardiac, renal, and cerebrovascular) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy.

Secondary outcomes

* To investigate the incidence and prevalence of FACEs with respect to Fabry specific treatment, Migalastat, ERT or no treatment.
* To describe FACEs in accordance with different geno- and phenotypic groups To investigate the incidence and time to a first fatal or non-fatal cardiac, renal and cerebrovascular clinical event, separated by each category.

Exploratory outcomes

- To describe disease progression with focus on organ involvement.

The study design is a retrospective clinical and paraclinical follow-up of the Danish National Fabry cohort in the period 01.01.2001-31.12.2022. Patient followed a structured yearly monitoring program as part of routine clincal care.

ELIGIBILITY:
Inclusion Criteria:

* Genetically-verified Fabry disease
* Age above or equal to 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients having been assessed for Fabry Disease in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first individual FACE since confirmed diagnosis (Composite endpoint) | 10 years post baseline
  Time to first FACE (cardiac, renal, and cerebrovascular) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy.
Time to first FACE after initiation of Migalastat treatment (Composite endpoint) | 5 years post baseline
  Time to first FACE (cardiac, renal, and cerebrovascular) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy.

SECONDARY OUTCOMES:
Time to first individual FACE since confirmed diagnosis (cardiac) | 10 years post baseline
  Time to first individual FACE (cardiac) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy.
Time to first individual FACE after initiation of Migalastat treatment (cardiac) | 5 years post baseline
  Time to first individual FACE (cardiac) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy.
Time to first individual FACE since confirmed diagnosis (renal) | 10 years post baseline
  Time to first individual FACE (renal) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy.
Time to first individual FACE after initiation of Migalastat treatment (renal) | 5 years post baseline
  Time to first individual FACE (renal) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy.
Time to first individual FACE after initiation of Migalastat treatment (cerebrovascular) | 5 years post baseline
  Time to first individual FACE (cerebrovascular) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy.
Time to first individual FACE since confirmed diagnosis (cerebrovascular) | 10 years post baseline
  Time to first individual FACE (cerebrovascular) with particular focus on Migalastat on clinical outcomes and treatment outcomes preceding Migalastat therapy.
Prevalence of FACE since confirmed diagnosis | 20 years post baseline
  The prevalence of FACEs since confirmed diagnosis
Prevalence of FACE after initiation of Fabry-specific treatment | 5 years post baseline
  The prevalence of FACEs after initiation of Fabry-specific treatment
Incidence of FACE since confirmed diagnosis | 20 years post baseline
  The incidence of FACEs since confirmed diagnosis
Incidence of FACE after initiation of Fabry-specific treatment | 5 years post baseline
  The incidence of FACEs after initiation of Fabry-specific treatment
Incidence of cardiac events since confirmed diagnosis | 20 years post baseline
  Incidence of cardiac, cerebrovascular, and renal clinical events separately by each specific category
Incidence of renal events since confirmed diagnosis | 20 years post baseline
  Incidence of cardiac, cerebrovascular, and renal clinical events separately by each specific category
Incidence of cerebrovascular events since confirmed diagnosis | 20 years post baseline
  Incidence of cardiac, cerebrovascular, and renal clinical events separately by each specific category
Incidence of cardiac events after initiation of Fabry-specific treatment | 5 years post baseline
  Incidence of cardiac, cerebrovascular, and renal clinical events separately by each specific category
Incidence of renal events after initiation of Fabry-specific treatment | 5 years post baseline
  Incidence of cardiac, cerebrovascular, and renal clinical events separately by each specific category
Incidence of cerebrovascular events after initiation of Fabry-specific treatment | 5 years post baseline
  Incidence of cardiac, cerebrovascular, and renal clinical events separately by each specific category
Annualized rate of change in eGFR by CKDEPI-formula since initiation of treatment | 20 years post baseline
  Annualized rate of change in eGFR based on the Chronic Kidney Disease Epidemiology Collaboration equation (eGFRCKD-EPI) over time to compare between Migalastat-treated, ERT, and untreated patients
Annualized rate of change in eGFR by CKDEPI-formula after initiation of Fabry-specific treatment | 5 years post baseline
  Annualized rate of change in eGFR based on the Chronic Kidney Disease Epidemiology Collaboration equation (eGFRCKD-EPI) over time to compare between Migalastat-treated, ERT, and untreated patients
Rapid renal progression of disease since confirmed diagnosis | 20 years post baseline
  Prevalence of clinically significant change in mGFR or eGFR defined as rapid progression (Using the KDIGO guidelines ie. sustained decline in GFR by 5 mL/min/1.73 m2/yr) since confirmed diagnosis.
Rapid renal progression of disease after initiation of Fabry-specific treatment | 5 years post baseline
  Prevalence of clinically significant change in mGFR or eGFR defined as rapid progression (Using the KDIGO guidelines ie. sustained decline in GFR by 5 mL/min/1.73 m2/yr) after initiation for Fabry-specific treatment.
Incidence of albuminuria since confirmed diagnosis | 20 years post baseline
  The incidence of albuminuria; defined as micro (> 30 mg/g creatinine) or macroalbuminuria (>300) by urinary albumin/creatinine ratio (ACR) or urinary 24 h protein excretion.
Incidence of albuminuria after initiation of Fabry-specific treatment | 5 years post baseline
  The incidence of albuminuria; defined as micro (> 30 mg/g creatinine) or macroalbuminuria (>300) by urinary albumin/creatinine ratio (ACR) or urinary 24 h protein excretion.
Prevalence of albuminuria since confirmed diagnosis | 20 years post baseline
  The prevalence of albuminuria; defined as micro (> 30 mg/g creatinine) or macroalbuminuria (>300) by urinary albumin/creatinine ratio (ACR) or urinary 24 h protein excretion.
Prevalence of albuminuria after initiation of Fabry-specific treatment | 5 years post baseline
  The prevalence of albuminuria; defined as micro (> 30 mg/g creatinine) or macroalbuminuria (>300) by urinary albumin/creatinine ratio (ACR) or urinary 24 h protein excretion.

OTHER OUTCOMES:
Organ-specific decline | 20 years post baseline
  Reflecting the montoring program of the annual clinical examinations and questionnaires of the Danish Fabry patients, the study will evaluate the organ-specific change prior to and after initiation of Fabry-specific treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Kistorp, MD, Ph.D, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to national legistlative restrictions, unrestricted access to individual participant data is not possible. However, data exchange will be possible upon reasonable request under the assurance of data-management in accordance with Danish law.

DOCUMENTS (2):
  • Study Protocol (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT06303466/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT06303466/SAP_001.pdf